CLINICAL TRIAL: NCT04507789
Title: Investigation of the Effectiveness of Exercise Training During Radiotherapy in Postoperative Breast Cancer
Brief Title: Exercise Therapy During Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Collaborators: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Damlagül AYDIN ÖZCAN, research assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-01
Record Dates: First submitted 2020-08-04; First posted 2020-08-11 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer; Exercise Therapy; Radiotherapy; Upper Extremity Problem
Keywords: Breast cancer; Exercise therapy; Radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise intervention group (Experimental): This group will be taken an exercise intervention during their radiotherapy programme.
  Interventions: Other: exercise intervention
- routine radiotherapy protocol (Active Comparator): This group will not be taken into an exercise intervention during their radiotherapy programme.
  Interventions: Other: routine radiotherapy protokol

INTERVENTIONS:
Other: exercise intervention — Exercise protocol will consist of the recommended special exercise sets for upper extremity problems on mastectomy patients. The upper extremity protocol has published in 2018 by Richmond and friends called prevention of musculoskeletal shoulder problems after breast cancer treatment UK-PROSPER protocol.this special protocol has unique exercise sets for to restore shoulder range of motion, to maintain good force level of upper extremity muscles and stretch exercises especially to the muscles around the radiotherapy area. Exercises will be done under the supervision of a specialized physiotherapist about upper extremity disorders.
  Arms: exercise intervention group
Other: routine radiotherapy protokol — This intervention is only an observation to patients during their routine radiotherapy protocol. There will be no exercise intervention for the upper extremity for the patient in this group.
  Arms: routine radiotherapy protocol

SUMMARY:
The main purpose of our study is to investigate the effects of exercise therapy on upper extremity functions in patients receiving radiotherapy to the axillary region after breast cancer surgery.

DETAILED DESCRIPTION:
Our study will take in place in radiation oncology clinic. In routine the patients which will receive axillary area radiotherapy will randomized into 2 groups will explained in study arms section later. There are papers explained about radiotherapy side effects to upper extremity functions. But there is lack of evidence about exercise therapy during radiotherapy protocol to cope with its side effects to upper extremity functions. In this study we will compare two groups upper extremity function related outcomes at the end of the radiotherapy sessions and also before and after results for two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients İn the age range of 18-65
* Receiving radiotherapy to the axillary region after surgery with breast cancer diagnosis

Exclusion Criteria:

* Radiotherapy area to contain only the chest wall
* Any orthopedic injury or trauma involving the upper extremity prior to or during the cancer diagnosis
* The presence of metastases in any area other than breast tissue

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-03-10 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
Upper extremity functional status of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  The subjective upper extremity functional status will assessed by The Disabilities of the Arm, Shoulder and Hand Score (DASH). This is 30 questions Questionnaire and 21 evaluate the person's difficulties during daily activities, 5 of them (pain, stiffness, tingling, weakness) and 4 of them evaluate work, sleep, social function and self-confidence. The person answers all questions according to the 5-point Likert system (1: no difficulty, 2: mild difficulty, 3: moderate difficulty, 4: extreme difficulty, 5: inability). A score of 0-100 is obtained from each section. As the score increases, the disability increases.
Shoulder joint range of motion (ROM) of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  Shoulder range of motion in flexion, abduction, internal rotation and external rotation will be evaluated by the standard goniometer. Total Active and passive degree of ROM will be evaluated in patient sitting position. Total ROM will record in degree value.
Hand Grip force measurement of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  Jamar hand dynamometer will be used for to evaluate gross hand grip force. While the patient is sitting with a back support in a comfortable seat, he will be asked to grasp the dynamometer with a gross grip at 90˚ flexion and compress it as strong as she can. 3 measurements will be made for both hands and the average of the values in kg will be recorded.

SECONDARY OUTCOMES:
Fear of movement, avoidance reaction of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  Tampa kinesiophobia ( fear of pain due to movement) scale will be used to evaluate the fear of movement degree. The survey has 17 question as a scale that is answered according to the 4-point Likert system. Total point will be between 17-68. As the score increases, the fear of movement increases.
Physical activity level of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  It will be evaluated by a short version of the International Physical Activity survey. The questionnaire consists of 7 questions and has open-ended questions for the physical activities to be filled in by the patient for the duration of activity and number of days.
Pain and sensory impairment of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  The McGill Pain short form scale will be used to evaluate patients sensory impairment. In the scale, 2 scores will be counted, first one is the total number of words defined by the person related to pain and sensation. Second score will be given by the patient to herself on visual analog scale in the range of 0-10. 10 means the worst pain while 0 is no pain.
Scapular dyskinesia of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  Lateral Slide Test method will be used to measure the scapular dyskinesia. In this method; While the patient is in a standing position the bottom corner of the scapula will be marked and the perpendicular length to the nearest vertebra will be measured with the help of tape for both scapulae. Then the same measurement will be repeated while the hands are at the waist and the hands are held in the 90˚ abduction position. The difference in scapula movement for both sides will be noted in cm.
Upper extremity kinesthesia and shoulder joint position sensation of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  While the patient's eyes closed and sitting on a chair, therapist's will be brought the shoulder range of motion to 90 degrees from the 0 degree start position. Meanwhile, angular value checks will be performed with an inclinometer fixed with velcro to mid-humeral area. A few seconds after the position is felt, the arm will be returned to the 0 degree start position. The patient will be asked to open his eyes and then he will be asked to actively bring his shoulder to the angle closest to the previous angle. Measurements will be made in 3 repetitions separately for the right and left sides and the degree differences will be determined for the sense of position and the average of the results will be taken.
Lymph edema evaluation of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  The lymph edema measurement will be made with a tape. The circumferential length around the arm will be made in every 5 cm from the distal tubercle to the shoulder. Studies have explained that a difference of up to 2 cm between both extremities can be considered normal and moderate and excessive lymph edema classification according to the difference in measurement. According to this staging, the severity of lymph edema in patients will be determined and recorded.
Life quality of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  It will be evaluated by EORTC QLQ-C30 (Cancer-specific quality of life index) . the questionnaire consists of 23 questions.The person answers all the questions according to the 4-point Likert system (1: none, 2: a little, 3: quite, 4: much). All sub scale points range between 0-100.
Breast cancer specific life quality of patients during radiotherapy protocol | ''day1 before radiotherapy session,'' ''after 6 week sessions of radiotherapy completed''
  It will be evaluated by EORTC QLQ-BR23 (Breast cancer-specific quality of life index). The questionnaire consists of 30 questions The person answers all the questions according to the 4-point Likert system (1: none, 2: a little, 3: quite, 4: much).All sub scale points range between 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: YAVUZ YAKUT, Study Chair — Professor; Güçlü Sezai Kılıçoğlu, Study Chair — assistant doctor
Locations (1):
- Dr. Abdurrahman Yurtaslan Onkoloji Hospital, Ankara, Yenimahalle, Turkey (Türkiye)